CLINICAL TRIAL: NCT05138718
Title: International Multicenter Trial on the Prognostic Value of Arterial 18F-FDG PET Imaging in Patients With History of Myocardial Infarction
Brief Title: FDG an Myocardial Infarction: The PIAF Trial
Acronym: PIAF
Status: Recruiting | Type: Observational
Sponsor: International Atomic Energy Agency (Other Government)
Responsible Party: Principal Investigator, Francesco Giammarile, Nuclear Medicine Physician, International Atomic Energy Agency
Other Study IDs: CRP13048
Record Dates: First submitted 2021-06-04; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: History of Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 18F-FDG PET/CT — Perform a 18F-FDG PET/CT to patients with history of myocardial infarction

SUMMARY:
In order to define distinct and reliable arterial 18Fluorodeoxyglucose (FDG) thresholds identifying patients at risk for cardiovascular events, patients with a history of myocardial infarction will be included in this international multicenter trial. Non-enhanced whole-body FDG PET/CT will be performed in all patients and the arterial FDG uptake in the carotid arteries as well as the aorta will be quantified by calculating different uptake parameters. In addition, FDG uptake in hematopoietic tissues (spleen, bone marrow), visceral adipose tissue (VAT) and different brain regions (e. g. amygdala) will be measured.

Furthermore, specific blood biomarkers including genetic biomarkers, which are linked to atherosclerotic disease with predictive power for future cardiovascular events, will be analyzed in a subgroup of patients. In part 2 of the trial, a 4-year follow-up period will be analyzed with a focus on the prediction of cardiovascular events (acute coronary syndrome, non-fatal ischemic stroke, ischemic cardiac death, other causes of death, coronary/vascular revascularization, new-onset of angina, symptomatic peripheral arterial disease and heart failure).

The predictive value of the arterial, hematopoietic and cerebral FDG uptake parameters as well as of the specific blood and genetic biomarkers will be determined.

DETAILED DESCRIPTION:
From a clinical perspective, atherosclerosis leading to arterial plaque rupture is one of the most important causes of death that still misses a personalized, reliable and quantitative assessment of risk. This is particularly true for patients who suffered from a non-fatal coronary syndrome, were recent studies described severe CVD event rates of up to 5 % per year despite the use of aggressive secondary prevention strategies.

While in previous clinical interventional trials inflammatory atherosclerotic activity was mainly determined by the surrogate marker high-sensitivity C-reactive protein, other studies have shown superiority of FDG PET/CT in the stratification of patients in high versus low risk groups, where risk in the highest (vs. lowest) TBR tertile was approximately 3-fold greater compared with what has been historically observed for the inflammatory blood biomarker, hsCRP. It is, thus, expected that imaging (vs. blood) biomarkers provide additional prognostic information that is more relevant to the artery wall per se, whereas currently used blood biomarkers carry information from vascular as well as nonvascular sources.

The current research aims at identifying distinct and reliable FDG PET threshold values, which specify the individual risk of a distinct patient. For this purpose, a well-designed and well-powered multicenter trial is needed.

Fundamentally, the research project aims at evaluating the prognostic value of arterial FDG PET/CT imaging of individuals with known cardiovascular disease (CVD). Specifically, we will:

* Test the hypothesis that the baseline measures of arterial inflammation (as assessed by FDG PET/CT) independently predict the risk of CVD events (as coronary death, myocardial infarction, coronary insufficiency, angina, ischemic stroke, hemorrhagic stroke, transient ischemic attack, peripheral artery disease, revascularization, or heart failure) in a large cohort of individuals with prior MI.
* Evaluate the incremental prognostic value of arterial inflammation (PET) over circulating blood biomarkers
* Evaluate the prognostic value of inflammation data derived from various arterial locations (e.g. aorta, carotids, or other locations) for their ability to predict severe cardiovascular events
* Identify cut-off values that indicate higher risk
* Evaluate the predicted value of specific brain uptake, hematopoietic tissue (spleen, bone marrow) and visceral adipose tissue on emerging CV events. Evaluate the added value of combining those uptake values with arterial uptake
* Evaluate the different established arterial FDG uptake parameters with regards to standardization and scanner type/variability
* Apply deep-learning algorithms for detection of organ/tissue interactions and CV event hypothesis generation
* Evaluate a subset of patients for inter-observer variability
* Evaluate the detection rate of incidental PET/CT findings in the study cohort (suspected malignancies, other diseases)
* Suggest novel diagnostic algorithms and clinical protocols accordingly
* Evaluate the prognostic value of additionally derived genetic markers.
* Specifically, we propose that patients with higher GRS have increased FDG PET/CT based inflammatory atherosclerotic activity and are prone to more MACE

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Patients 18-80 years of age
* Patients with documented myocardial infarction > 90 days before study inclusion
* Clinically stable at the time of screening and able to tolerate the study procedure
* Female patients must not be pregnant at the time of FDG PET/CT imaging
* Patients included in other clinical trials could be included, provided this complies with specific local and research center requirements
* If after 6 months of patient recruitment it is foreseeable that the target number of patients will not be reached, patients who undergo FDG PET/CT imaging for cancer screening or surveillance can be included, provided that they have no evidence of an active malignancy on the scan or other exclusion criteria as listed below at study entry, including recent radio- and / or chemotherapy (≥ 12 months before the FDG PET/CT)

Exclusion Criteria:

* Severe congestive heart failure (class III or IV according to NYHA, or pulmonary edema)
* Extra-cardiac illness that is expected to limit survival to less than 4-5 years; e. g. oxygen-dependent chronic obstructive pulmonary disease, active hepatitis or severe hepatic dysfunction, severe renal disease, active cancer
* Patients with chronic use of anti-inflammatory medication (except NSAIDs and inhaled corticosteroids)
* Patients with Diabetes Type I
* Insulin-dependent or uncontrolled Diabetes Type II (as HbA1C>7.5)
* Withdrawal of Informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients 18-80 years of age
  * Patients with documented myocardial infarction > 90 days before study inclusion
  * Clinically stable at the time of screening and able to tolerate the study procedure
Sampling Method: Non-Probability Sample
Enrollment: 2041 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular events | 4 to 5 years follow-up period
  Cardiovascular events considered will be: coronary death, myocardial infarction, coronary insufficiency/acute coronary syndrome, angina, ischemic stroke, hemorrhagic stroke, transient ischemic attack, peripheral artery disease, revascularization, or heart failure

SECONDARY OUTCOMES:
Other cardiovascular events | 4 to 5 years follow-up period
  coronary/vascular revascularization, new-onset of angina, symptomatic peripheral arterial disease and heart failure
All-causes of death | 4 to 5 years follow-up period
  All-causes of death

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Giammarile, MD, PhD, Study Director — International Atomic Energy Agency
Locations (1):
- Massachusetts General Hospital, Havard Medical School, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iwatsuka R, Matsue Y, Yonetsu T, O'uchi T, Matsumura A, Hashimoto Y, Hirao K. Arterial inflammation measured by 18F-FDG-PET-CT to predict coronary events in older subjects. Atherosclerosis. 2018 Jan;268:49-54. doi: 10.1016/j.atherosclerosis.2017.11.016. Epub 2017 Nov 21. PMID 29175654
- [Background] Figueroa AL, Abdelbaky A, Truong QA, Corsini E, MacNabb MH, Lavender ZR, Lawler MA, Grinspoon SK, Brady TJ, Nasir K, Hoffmann U, Tawakol A. Measurement of arterial activity on routine FDG PET/CT images improves prediction of risk of future CV events. JACC Cardiovasc Imaging. 2013 Dec;6(12):1250-9. doi: 10.1016/j.jcmg.2013.08.006. Epub 2013 Oct 23. PMID 24269261
- [Background] Duivenvoorden R, Mani V, Woodward M, Kallend D, Suchankova G, Fuster V, Rudd JHF, Tawakol A, Farkouh ME, Fayad ZA. Relationship of serum inflammatory biomarkers with plaque inflammation assessed by FDG PET/CT: the dal-PLAQUE study. JACC Cardiovasc Imaging. 2013 Oct;6(10):1087-1094. doi: 10.1016/j.jcmg.2013.03.009. PMID 24135322
- [Background] Nitta Y, Tahara N, Tahara A, Honda A, Kodama N, Mizoguchi M, Kaida H, Ishibashi M, Hayabuchi N, Ikeda H, Yamagishi S, Imaizumi T. Pioglitazone decreases coronary artery inflammation in impaired glucose tolerance and diabetes mellitus: evaluation by FDG-PET/CT imaging. JACC Cardiovasc Imaging. 2013 Nov;6(11):1172-82. doi: 10.1016/j.jcmg.2013.09.004. PMID 24229770
- [Background] Noh TS, Moon SH, Cho YS, Hong SP, Lee EJ, Choi JY, Kim BT, Lee KH. Relation of carotid artery 18F-FDG uptake to C-reactive protein and Framingham risk score in a large cohort of asymptomatic adults. J Nucl Med. 2013 Dec;54(12):2070-6. doi: 10.2967/jnumed.113.119602. Epub 2013 Oct 31. PMID 24179183
- [Background] Hetterich H, Rominger A, Walter L, Habs M, Volpers S, Hacker M, Reiser MF, Bartenstein P, Saam T. Natural history of atherosclerotic disease progression as assessed by (18)F-FDG PET/CT. Int J Cardiovasc Imaging. 2016 Jan;32(1):49-59. doi: 10.1007/s10554-015-0660-8. Epub 2015 Apr 22. PMID 25898891
- [Result] D'Agostino RB Sr, Vasan RS, Pencina MJ, Wolf PA, Cobain M, Massaro JM, Kannel WB. General cardiovascular risk profile for use in primary care: the Framingham Heart Study. Circulation. 2008 Feb 12;117(6):743-53. doi: 10.1161/CIRCULATIONAHA.107.699579. Epub 2008 Jan 22. PMID 18212285